CLINICAL TRIAL: NCT00002637
Title: PHASE I/II STUDY OF IMMUNIZATION WITH MHC CLASS I MATCHED ALLOGENEIC HUMAN PROSTATIC CARCINOMA CELLS ENGINEERED TO SECRETE INTERLEUKIN-2 AND INTERFERON-GAMMA
Brief Title: Biological Therapy in Treating Patients With Prostate Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Purpose: Treatment
Other Study IDs: 94-134; CDR0000064100 (Registry Identifier: PDQ (Physician Data Query)); NCI-V95-0629
Record Dates: First submitted 1999-11-01; First posted 2004-06-10 (Estimated); Last update posted 2013-06-25 (Estimated); Status verified 2013-06

CONDITIONS: Prostate Cancer
Keywords: recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — aldesleukin; Interferon-gamma

INTERVENTIONS:
Biological: aldesleukin
Biological: gene-modified tumor cell vaccine therapy
Biological: recombinant interferon gamma

SUMMARY:
RATIONALE: Interleukin-2 may stimulate a person's white blood cells including natural killer cells to kill prostate cancer cells. Interferon gamma may interfere with the growth of the cancer cells. Combining interferon gamma with interleukin-2 may be a more effective treatment for prostate cancer.

PURPOSE: Phase I/II trial to study the effectiveness of biological therapy using interleukin-2 and interferon gamma in treating patients with advanced prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the safety of immunization with HLA class I-matched allogeneic human prostate carcinoma cells genetically engineered to secrete interleukin-2 and interferon gamma in patients with prostate carcinoma. II. Evaluate the antitumor effects of this treatment as assessed by post-therapy declines in PSA. III. Evaluate the induction of cellular and humoral immunity in vivo with this treatment.

OUTLINE: Tumor Cell Vaccine Therapy. Immunization with irradiated, MHC class I-matched allogeneic human prostate carcinoma cells, LNCaP cells, engineered to secrete approximately 58 ng/24 hr/million cells of interleukin-2 (IL-2) and approximately 0.72 U/24 hr/million cells of interferon gamma (IFN-G).

PROJECTED ACCRUAL: Up to 12 patients will be entered on the Phase I study; accrual will continue to a total of 25 patients treated at the MTD (Phase II). Accrual is expected to require 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed prostate carcinoma For Phase I: progressive, androgen-independent disease required, i.e.: Elevated PSA despite castrate testosterone levels (below 50 ng/dl) documented on 3 successive occasions For Phase II: progressive disease after surgery or radiotherapy without prior hormonal therapy also eligible HLA-A1- or HLA-A2-positive disease required Measurable or evaluable disease required No active CNS metastases

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 70-100% Life expectancy: At least 12 weeks Hematopoietic: WBC greater than 3,000 Absolute lymphocytes greater than 1,000 Platelets greater than 100,000 Hb at least 9 g/dl Hepatic: Bilirubin less than 2.0 mg/dl OR SGOT less than 2 x ULN Renal: Creatinine no greater than 2.0 mg/dl OR Creatinine clearance at least 40 ml/min Cardiovascular: No NYHA class III/IV status Pulmonary: No severe debilitating pulmonary disease Other: No active infection requiring antibiotics Not HIV positive No history of hypersensitivity to interferon gamma or other vaccine component No serious intercurrent medical illness

PRIOR CONCURRENT THERAPY: Recovered from toxicity of any prior therapy Biologic therapy: No prior autologous or allogeneic tumor vaccines No concurrent other immunotherapy Chemotherapy: At least 4 weeks since chemotherapy No concurrent chemotherapy Endocrine therapy: Flutamide discontinued and subsequent progression prior to entry 3 consecutive rising PSA values at least 2 weeks apart No concurrent corticosteroids (except for life-threatening conditions) Medical hormonal therapy to maintain castrate testosterone levels required in the absence of orchiectomy Radiotherapy: At least 4 weeks since radiotherapy No concurrent radiotherapy Surgery: Prior surgery allowed

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 1995-01; Primary Completion 2001-02 (Actual); Study Completion 2001-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Slovin, MD, PhD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States